CLINICAL TRIAL: NCT04530123
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 2 Dose-Ranging Study to Evaluate the Efficacy and Safety of TAK-101 for the Prevention of Gluten-Specific T Cell Activation in Subjects With Celiac Disease on a Gluten-Free Diet
Brief Title: Dose-Ranging Study of the Efficacy and Safety of TAK-101 for Prevention of Gluten-Specific T Cell Activation in Participants With Celiac Disease on a Gluten-Free Diet
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TAK-101-2001; U1111-1253-8169 (Registry Identifier: World Health Organization)
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Celiac Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Celiac Disease | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1, Group A: Placebo + Placebo + TAK-101 25 µg/kg GE (Experimental): Following a single-day 3 gram (g) oral run-in gluten challenge, participants will receive TAK-101 placebo-matching intravenous (IV) infusion dose, once each on Days 1 and 8, followed by 12 g/day gluten for 3 days followed by 6 g/day gluten for 3 days starting at Week 2. Participants will then undergo single-day 3 g gluten challenges at Weeks 8, 14, and 20. A third IV infusion dose of TAK-101 25 microgram per kilogram (µg/kg) GE will be given 23 weeks after the second dose at approximately Week 24.
  Interventions: Drug: Placebo; Drug: TAK-101; Dietary Supplement: Gluten
- Cohort 1, Group B: TAK-101 25 µg/kg GE + Placebo + TAK-101 25 µg/kg GE (Experimental): Following a single-day 3 g oral run-in gluten challenge, participants will receive TAK-101 25 µg/kg, IV infusion once on Day 1 followed by TAK-101 placebo-matching IV infusion, once on Day 8, followed by 12 g/day gluten for 3 days followed by 6 g/day gluten for 3 days starting at Week 2. Participants will then undergo single-day 3 g gluten challenges at Weeks 8, 14, and 20. A third IV infusion dose of TAK-101 25 µg/kg GE will be given 23 weeks after the second dose at approximately Week 24.
  Interventions: Drug: Placebo; Drug: TAK-101; Dietary Supplement: Gluten
- Cohort 1, Group C: TAK-101 25 µg/kg GE + TAK-101 25 µg/kg GE + TAK-101 25 µg/kg GE (Experimental): Following a single-day 3 g oral run-in gluten challenge, participants will receive TAK-101 25 µg/kg GE IV infusion, once each on Days 1 and 8, followed by 12 g/day gluten for 3 days followed by 6 g/day gluten for 3 days starting at Week 2. Participants will then undergo single-day 3 g gluten challenges at Weeks 8, 14, and 20. A third IV infusion dose of TAK-101 25 µg/kg GE will be given 23 weeks after the second dose at approximately Week 24.
  Interventions: Drug: TAK-101; Dietary Supplement: Gluten
- Cohort 2, Group A: Placebo + Placebo + TAK-101 25 µg/kg GE (Experimental): Following a single-day 3 g oral run-in gluten challenge, participants will receive TAK-101 placebo-matching IV infusion, once each on Days 1 and 8, followed by 12 g/day gluten for 3 days followed by 6 g/day gluten for 3 days starting at Week 2. Participants will then undergo single-day 3 g gluten challenges at Weeks 8, 14, and 20. A third IV infusion dose of TAK-101 25 µg/kg GE will be given 23 weeks after the second dose at approximately Week 24. Cohort 2 would start based on the results of Cohort 1.
  Interventions: Drug: Placebo; Drug: TAK-101; Dietary Supplement: Gluten
- Cohort 2, Group D: TAK-101 50 µg/kg GE + TAK-101 50 µg/kg GE+ TAK-101 50 µg/kg GE (Experimental): Following a single-day 3 g oral run-in gluten challenge, participants will receive TAK-101 50 µg/kg GE IV infusion, once each on Days 1 and 8, followed by 12 g/day gluten for 3 days followed by 6 g/day gluten for 3 days starting at Week 2. Participants will then undergo single-day 3 g gluten challenges at Weeks 8, 14, and 20. A third IV infusion dose of TAK-101 50 µg/kg GE will be given 23 weeks after the second dose at approximately Week 24. Cohort 2 would start based on the results of Cohort 1.
  Interventions: Drug: TAK-101; Dietary Supplement: Gluten
- Cohort 2, Group E: Placebo + Placebo + TAK-101 12.5 µg/kg GE (Experimental): Following a single-day 3 g oral run-in gluten challenge, participants will receive TAK-101 placebo-matching IV infusion, once each on Days 1 and 8, followed by 12 g/day gluten for 3 days followed by 6 g/day gluten for 3 days starting at Week 2. Participants will then undergo single-day 3 g gluten challenges at Weeks 8, 14, and 20. A third IV infusion dose of TAK-101 12.5 µg/kg GE will be given 23 weeks after the second dose at approximately Week 24. Cohort 2 would start based on the results of Cohort 1. This group would be opened only if it is decided not to open Cohort 2 at the 50 µg/kg GE dose level.
  Interventions: Drug: Placebo; Drug: TAK-101; Dietary Supplement: Gluten
- Cohort 2, Group F: TAK-101 12.5 µg/kg GE + TAK-101 12.5 µg/kg GE + TAK-101 12.5 µg/kg GE (Experimental): Following a single-day 3 g oral run-in gluten challenge, participants will receive TAK-101 12.5 µg/kg GE IV infusion, once each on Days 1 and 8, followed by 12 g/day gluten for 3 days followed by 6 g/day gluten for 3 days starting at Week 2. Participants will then undergo single-day 3 g gluten challenges at Weeks 8, 14, and 20. A third IV infusion dose of TAK-101 12.5 µg/kg GE will be given 23 weeks after the second dose at approximately Week 24. Cohort 2 would start based on the results of Cohort 1.
  Interventions: Drug: TAK-101; Dietary Supplement: Gluten

INTERVENTIONS:
Drug: Placebo — TAK-101 placebo-matching intravenous infusion
  Arms: Cohort 1, Group A: Placebo + Placebo + TAK-101 25 µg/kg GE; Cohort 1, Group B: TAK-101 25 µg/kg GE + Placebo + TAK-101 25 µg/kg GE; Cohort 2, Group A: Placebo + Placebo + TAK-101 25 µg/kg GE; Cohort 2, Group E: Placebo + Placebo + TAK-101 12.5 µg/kg GE
Drug: TAK-101 — TAK 101 intravenous infusion
Dietary Supplement: Gluten — Powder form (vital wheat gluten)

SUMMARY:
The main aim of the study is to assess if TAK-101 can reduce gluten related symptoms and immune activation in adult participants with celiac disease (CeD) on a gluten-free diet (GFD).

Participants will receive TAK-101 and/or placebo through the vein on Day 1 and Day 8. All participants will receive active treatment at Week 24.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-101. TAK-101 is being tested to treat people who have celiac disease. The study has 2 cohorts planned. Cohort 1 has 1 dose level and the Cohort 2 may include 1 or 2 additional dose levels, depending on safety, tolerability, and activity observed in Cohort 1. Dosing in the Cohort 2 will be based on data from Cohort 1.

The study will enroll approximately 90 patients. In Cohort 1, approximately 45 participants will be randomly assigned in 1:2:2 ratio in one of the three arm groups which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need). Eligible participants in Cohort 1 will receive:

* Group A: 2 infusion doses of placebo, 1 infusion dose on Day 1 and 1 infusion dose on Day 8, followed by 1 infusion dose of 25 micrograms per kilogram (µg/kg) Gluten Epitopes (GE) TAK-101 at Week 24.
* Group B: 1 infusion dose of 25 µg/kg GE TAK-101 on Day 1 followed by 1 infusion dose of placebo on Day 8, followed by 1 infusion dose of 25 µg/kg GE TAK-101 at Week 24.
* Group C: 2 infusion doses of 25 µg/kg GE TAK-101, 1 infusion dose on Day 1 and 1 infusion dose on Day 8, followed by 1 infusion dose of 25 µg/kg GE TAK-101 at Week 24.

If it is deemed appropriate to enroll both the TAK-101 50 µg/kg GE and the 12.5 µg/kg GE dose levels in Cohort 2, approximately 45 participants may be randomly assigned in 1:2:2 ratio in Cohort 2 to receive:

* Group A: Two infusion doses of placebo, 1 infusion dose on Day 1 and 1 infusion dose on Day 8, followed by 1 infusion dose of 25 µg/kg GE TAK-101 at Week 24.
* Group D: Two infusion doses of 50 µg/kg GE TAK-101, 1 infusion dose on Day 1 and 1 infusion dose on Day 8, followed by 1 infusion dose of 50 µg/kg GE TAK-101 at Week 24.
* Group F: Two infusion doses of 12.5 µg/kg GE TAK-101, 1 infusion dose on Day 1 and 1 infusion dose on Day 8, followed by 1 infusion dose of 12.5 µg/kg GE TAK-101 at Week 24.

If it is decided not to open the second cohort at the 50 µg/kg GE dose level and if 1 2.5 µg/kg GE dose is recommended to be tested by the independent data monitoring committee (IDMC), approximately 27 participants will be randomly assigned in 1:2 ratio to receive:

* Group E: Two infusion doses of placebo, 1 infusion dose on Day 1 and 1 infusion dose on Day 8, followed by 1 infusion dose of 12.5 µg/kg GE TAK-101 at Week 24.
* Group F: Two infusion doses of 12.5 µg/kg GE TAK-101, 1 infusion dose on Day 1 and 1 infusion dose on Day 8, followed by 1 infusion dose of 12.5 µg/kg TAK-101 at Week 24.

This trial will be conducted globally. The overall time to participate in this study is approximately 34 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone OR plus a final visit after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-confirmed CeD that is well-controlled, defined as mild or with no ongoing signs or symptoms felt to be related to active CeD and with immunoglobulin A (IgA) tissue transglutaminase (tTG) <2 × upper limit of normal (ULN) and IgG deamidated gliadin peptide (DGP) <3 × ULN.

   Note: Participants may be retested for IgA tTG and IgG DGP to meet eligibility criteria at the discretion of the investigator. Intermittent symptoms would not exclude participants from participation as long as symptoms are generally well controlled in the opinion of the investigator, and as long as symptoms are back to baseline for 2 weeks before the run-in gluten challenge.
2. Must be able to maintain a gluten-free diet (GFD) for ≥6 months.
3. Must be HLA-DQ2.5 and/or HLA-DQ8 positive during screening laboratory testing.

Exclusion Criteria:

1. Has received any investigational compound within 12 weeks (84 days) or 5 half-lives, whichever is longer, before signing of the informed consent form (ICF).
2. Has received TAK-101 in a previous clinical study.
3. Has presence of other inflammatory gastrointestinal (GI) disorders or systemic autoimmune diseases, that either have the potential to cause persistent GI symptoms similar to CeD or are not well controlled without the use of excluded medications.

   * Examples of conditions that are exclusionary include: inflammatory bowel disease, eosinophilic gastroenteritis or colitis, and microscopic colitis requiring treatment in the 6 months before screening.
   * Examples of conditions that may be permissible after discussion with the medical monitor/or sponsor include: systemic autoimmune disease such as scleroderma, psoriatic or rheumatoid arthritis, lupus that is stable and without GI involvement, well controlled autoimmune thyroid disease, well controlled type 1 diabetes or proton pump inhibitor -responsive eosinophilic esophagitis in symptomatic and histologically confirmed remission.
4. Has known or suspected refractory CeD or ulcerative jejunitis.
5. Has known or suspected allergy to wheat, such as hypersensitivity and/or anaphylaxis including wheat-dependent-exercise induced anaphylaxis (WDEIA). If there is a possible history of urticaria, angioedema, or anaphylaxis to wheat, investigators should perform testing for wheat anti-Immunoglobulin (anti-IgE) antibodies or refer to an allergist for evaluation prior to enrollment to rule out any of these allergies.
6. Ongoing systemic immunosuppressant, systemic (oral or IV) corticosteroid treatment, or has received treatment with systemic immunosuppressants or corticosteroids in the 12 weeks before run-in gluten challenge.
7. Has known or suspected clinically significant liver disease or positive test result for hepatitis B or C.
8. Has intolerable symptoms after the run-in gluten challenge and is unwilling to undergo subsequent post treatment gluten challenges.
9. Has known allergy to or intolerance of TAK-101 or any of its ingredients or excipients. Also, any subject with a symptomatic allergic reaction that is confirmed by laboratory serology such as elevated tryptase levels following the administration of TAK-101 will be excluded from future dosing.
10. Has a current diagnosis of active malignancy or malignancy diagnosed in the 5 years prior to screening or is receiving ongoing treatment for malignancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-01-08 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Interferon-gamma Spot Forming Units (IFN-γ SFUs) in Human Leukocyte Antigens Density Quotient (HLA-DQ2.5-positive) Participants Based on Results of a Gliadin-Specific Enzyme-Linked Immunospot (ELISpot) Assay | Baseline (Day 15, or Day 1 in the absence of Day 15) to Week 3 (Day 20)
  IFN-γ SFUs will be measured based on results of a gliadin-specific ELISpot assay using gluten-specific T cells which will be isolated from blood.

SECONDARY OUTCOMES:
Percentage of Participants Experiencing at Least One Adverse Event (AE) and Adverse Events of Special Interest (AESIs) | From the first IV dose up to 30 days after last IV dose (Up to Week 28)
  An AE is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a markedly abnormal physical examination finding, vital sign value, laboratory test value), symptom, or disease temporally associated with the use of a drug whether or not it is considered related to the drug. An AESI (serious or nonserious) is one of scientific and medical concern specific to the compound or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor may be appropriate.
Change From Run-in (Visit 2) to Weeks 8, 14, and 20 in the Pre- to Post-gluten Challenge Change of the 3-day Average Nausea Severity Score as Measured in Celiac Disease Symptom Diary (CDSD) | Run-in (Visit 2), Weeks 8, 14, and 20
  The CDSD version 2.1 is an 8-item, self-administered questionnaire that evaluates the celiac disease (CeD) symptoms using 5-point Likert-type scales, where lower score indicating no symptoms and higher score indicating severe symptoms for all items except for frequency questions relating to stool counts, diarrhea, and vomiting frequency. The scores from the past 3 days with a 24-hour recall period will be averaged. For Weeks 8, 14, and 20, it is calculated as the average of the available daily scores recorded in the 3 days prior and after the respective gluten challenge.
Change From Run-in (Visit 2) to Weeks 8,14, and 20 in the Pre- to Post-gluten Challenge Change in CDSD 3-day Peak Nausea Severity Score | Run-in (Visit 2), Weeks 8, 14, and 20
  The CDSD version 2.1 is an 8-item, self-administered questionnaire that evaluates the CeD symptoms using 5-point Likert-type scales, where lower score indicating no symptoms and higher score indicating severe symptoms for all items except for frequency questions relating to stool counts, diarrhea, and vomiting frequency. The scores from the past 3 days with a 24-hour recall period will be averaged. Peak score is the highest score in the 3 days prior and following gluten challenge at Weeks 8, 14, and 20.
Change From Run-in (Visit 2) to Weeks 8, 14, and 20 in the Pre- to Post-gluten Challenge Change in Weekly Gastrointestinal (GI) Symptom Severity Score | Run-in (Visit 2), Weeks 8, 14, and 20
  The CDSD version 2.1 is an 8-item, self-administered questionnaire that evaluates the CeD symptoms using 5-point Likert-type scales, where lower score indicating no symptoms and higher score indicating severe symptoms for all items except for frequency questions relating to stool counts, diarrhea, and vomiting frequency. GI symptom severity score ranges from 0 to 20 with higher score indicating more severe disease.
Fold Change in Plasma Interleukin-2 (IL-2) from Run-in (Visit 2) to Day 15, and Weeks 8, 14, and 20 | Pre-/post-gluten challenge at Run-in (Visit 2), Day 15, and Weeks 8, 14, and 20
  The pre-/post-gluten challenge fold change in plasma IL-2 from Run-in (Visit 2) to Day 15, and Weeks 8, 14, and 20 will be compared.
Fold Change in Plasma IL-2 at Specified Time Points | Pre-/post-gluten challenge at Run-in (Visit 2), Day 15, and Weeks 8, 14, and 20
  The pre-/post-gluten challenge fold change in plasma IL-2 at each of the time points will be compared.
Plasma Concentration of TAK-101 After Each Dose | Predose and postdose at Weeks 0, 1 and 24
Serum Concentration of Antidrug Antibody (ADAs) to Various Doses of TAK-101 | Predose at Week 1 and before gluten challenge at Weeks 2, 14, 20, and 24
  ADA includes deamidated gliadin peptide- immunoglobulin G (DGP- IgG).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (48):
- United States (26):
  - One of a Kind Clinical Research Center LLC, Scottsdale, Arizona
  - Gastroenterology and Liver Institute, Escondido, California
  - Cadena Care Institute, Inc., Poway, California
  - Asthma and Allergy Associates, PC, Colorado Springs, Colorado
  - GCP Clinical Research, LLC, Tampa, Florida
  - Agile Clinical Research Trials, Atlanta, Georgia
  - Lemah Creek Clinical Research, Burr Ridge, Illinois
  - Gastroenterology Associates, PA, Rockford, Illinois
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Berkshire Medical Center, New Albany, Indiana
  - Gastroenterology Health Partners, PLLC, New Albany, Indiana
  - Boston Specialists, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Berkshire Medical Center, Inc., Pittsfield, Massachusetts
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Wellness Clinical Research, Chesterfield, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Basil Clinical, Inwood, New York
  - Mount Sinai, New York, New York
  - Columbia University Medical Center. New York Presbyterian Hospital, New York, New York
  - East Carolina Gastroenterology, PA, Jacksonville, North Carolina
  - GI Alliance-Rhode Island, Providence, Rhode Island
  - Amel Med LLC, Georgetown, Texas
  - Care Access Research - Salt Lake City, Ogden, Utah
- Australia (9):
  - Royal Melbourne Hospital, Parkville, AU
  - Emeritus Research, Sydney, Botany, NS
  - Coral Sea Clinical Research Institute, North Mackay, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Emeritus Research, Melbourne, Camberwell, Victoria
  - The Northern Hospital, Epping, Victoria
  - St John of God Midland, Midland, Western Australia
  - St Vincent's Hospital Melbourne, Fitzroy
  - Mater Hospital Brisbane, South Brisbane
- Canada (5):
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton, Alberta
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - McMaster University, Hamilton, Ontario
  - Scott Shulman Medicine Professional Corporation, North Bay, Ontario
  - DIEX Recherche Quebec Inc., Québec, Quebec
- New Zealand (8):
  - Silverdale Medical, Silverdale, Auckland
  - Optimal Clinical Trials - North, Auckland, AU
  - Southern Clinical Trials Totara, New Lynn, AU
  - Momentum Clinical Research Dunedin, Dunedin, OT
  - P3 Research Limited (Wellington), Wellington, OT
  - Capital, Coast and Hutt Valley - Wellington Regional Hospital, Boulcott, WG
  - Lakeland Clinical Trials Wellington, Upper Hutt, WG
  - Optimal Clinical Trials - Central, Grafton

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/5f8339975a55120029fe7d9c?idFilter=%5B%22TAK-079-1004%22%2C%22TAK-101-2001%22%5D